CLINICAL TRIAL: NCT02612805
Title: Effects of Two Models of Physical Training in Aquatic Environment in Control of Type 2 Diabetes - A Controled Randomized Clinical Trial: The Diabetes and Aquatic Training Study (DATS)
Brief Title: The Diabetes and Aquatic Training Study (DATS)
Acronym: DATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0380
Record Dates: First submitted 2015-11-11; First posted 2015-11-24 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic training group (Experimental): This group perform aerobic hydrogymnastics.
  Interventions: Other: Aerobic training
- Combined training group (Active Comparator): This group perform combined hydrogymnastics.
  Interventions: Other: Combined training
- Training placebo (Placebo Comparator): This group perform stretching and relaxation in aquatic environment.
  Interventions: Other: Training placebo

INTERVENTIONS:
Other: Aerobic training — Total duration of exercise sessions: 56 minutes (3 minutes of warming - 50 minutes of main part - 3 minutes of stretching); Method of training: Aerobic continuous in aquatic environment; Modality: Hydrogymnastics; Weekly frequency: 3; Intensity: 85% to 100% of the anaerobic threshold during the intervention.
  Other Names: Aquatic aerobic training
  Arms: Aerobic training group
Other: Combined training — Total duration of exercise sessions: 56 minutes (3 minutes of warming - 50 minutes of main part - 3 minutes of stretching); Method of training: Aerobic more resistance training.
  Aerobic component (between 30 and 40 minutes of the sessions): Method: Aerobic continuous in aquatic environment; Modality: Hydrogymnastics; Weekly frequency: 3; Intensity: 85% to 100% of the anaerobic threshold during the intervention.
  Resistance component (Between 10 and 20 minutes of the sessions): Method: Multiple sets (2 to 4 sets of 30 to 15 seconds) in aquatic environment; Modality: Hydrogymnastics; Weekly frequency: 3; Intensity: Maximum execution speed.
  Other Names: Aquatic combined training
  Arms: Combined training group
Other: Training placebo — Total duration of exercise sessions: 56 minutes (3 minutes of warming - 50 minutes of main part - 3 minutes of stretching); Activities performed in main part: Stretching and relaxation in aquatic environment.
  Other Names: Control procedure
  Arms: Training placebo

SUMMARY:
This study evaluates the effects of the combined exercise training (aerobic more resistance) and of the aerobic exercise training isolated compared to control group, which performed only stretching and relaxation, in the treatment of type 2 diabetes (T2DM). The two exercise interventions and the control procedure are performed in aquatic environment.

DETAILED DESCRIPTION:
The fact that aquatic training can provide similar benefits to land training has important clinical implications, because the aquatic environment provides some interesting advantages to this population, such as no impact on walking and running in deep water or reduced, as in water-based exercises. This minor impact and consequent reduced chance of injury allows consider the aquatic environment favorable to the principle of continuity with progression of physiological stimuli and metabolic benefits.

From these peculiarities of the training in aquatic environment, and of the association between T2DM with obesity and hypertension, conditions that create difficulties for individuals performing exercise supporting their own body mass and need both benefits from aerobic and resistance training, is believed to be necessary to carry out physical training programs of the same duration, differing in training mode (aerobic or combined) in the aquatic environment in order to answer of in a adequated duration of training, the diabetes control through training differs between the different mode of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* Be under medical treatment with oral hypoglycemic agents and / or insulin;
* Not engaged in regular exercise (regular exercise was defined as performing any type of physical training for at least 20 minutes three or more days a week).

Exclusion Criteria:

* Severe autonomic neuropathy;
* Severe nonproliferative and proliferative diabetic retinopathy;
* Decompensated heart failure;
* Limb amputations;
* Severe foot injuries;
* Chronic renal failure (Modification Diet in Renal Disease-MDRD, Glomerular Filtration Rate-GFR < 30 ml/min);
* Body mass index (BMI) > 45.0 kg/m2;
* Any muscle or joint impairment which prevented individuals from engaging in physical exercise.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in levels of glycated hemoglobin | Change from Baseline levels of glycated hemoglobin at 15-weeks.

SECONDARY OUTCOMES:
Fasting plasma glucose. | At baseline and after a 15-week period.
Fasting insulin. | At baseline and after a 15-week period.
Insulin-resistance index (HOMA-IR). | At baseline and after a 15-week period.
Total cholesterol. | At baseline and after a 15-week period.
high density lipoprotein. | At baseline and after a 15-week period.
Low density lipoprotein. | At baseline and after a 15-week period.
Triglycerides. | At baseline and after a 15-week period.
Renin | At baseline and after a 15-week period.
High sensitive C-reactive protein. | At baseline and after a 15-week period.
Total testosterone. | At baseline and after a 15-week period.
Cortisol | At baseline and after a 15-week period.
Testosterone/cortisol ratio. | At baseline and after a 15-week period.
Peak oxygen uptake. | At baseline and after a 15-week period.
Oxygen uptake at the second ventilatory threshold. | At baseline and after a 15-week period.
Percentage of oxygen consumption in the second ventilatory threshold from the peak oxygen uptake. | At baseline and after a 15-week period.
Systolic blood pressure. | At baseline and after a 15-week period.
Diastolic blood pressure | At baseline and after a 15-week period.
Heart rate at rest. | At baseline and after a 15-week period.
Maximum dynamic muscle strength (1RM) in the knees extension exercise. | At baseline and after a 15-week period.
  The test is characterized by greater load that can be supported in a single execution of knees extension exercise.
Maximum dynamic muscle strength (1RM) in the elbows flexion exercise. | At baseline and after a 15-week period.
  The test is characterized by greater load that can be supported in a single execution of elbows flexion exercise.
Resistant dynamic muscle strength (maximal repetitions) in the knees extension exercise. | At baseline and after a 15-week period.
  To determine the resistant dynamic muscle strength, it was considered the number of repetitions performed at 60% of 1RM, following a pace and breadth of pre-established execution. In the post-training evaluation, we used the load of 60% of 1RM test performed in the pre-training.
Resistant dynamic muscle strength (maximal repetitions) in the elbows flexion exercise. | At baseline and after a 15-week period.
  To determine the resistant dynamic muscle strength, it was considered the number of repetitions performed at 60% of 1RM, following a pace and breadth of pre-established execution. In the post-training evaluation, we used the load of 60% of 1RM test performed in the pre-training.
Timed up and go test performed at the usual speed. | At baseline and after a 15-week period.
Timed up and go test performed at the maximal speed. | At baseline and after a 15-week period.
Sitting-rising test (SRT). | At baseline and after a 15-week period.
  The SRT basically consists in the quantification of the number of support (hands and/or knees, or hands or forearms on knees) one utilizes in order to sit and to rise from the floor.
Overall quality of life and in physical, psychological, social relationships and environment domains, evaluated by instrument of World Health Organization (WHOQOL). | At baseline and after a 15-week period.
  To evaluate the quality of life we used the WHOQOL-brief instrument. This instrument is self-applicable, cross-cultural, translated and validated for Portuguese, consisting of 26 questions. Its score ranges from zero to 100 points, divided into the physical, psychological, social relationships and environment, as well as an assessment of the overall quality of life.
Depressive symptoms, evaluated by Depression Inventory Patient Health Questionnarie (PHQ-9) | At baseline and after a 15-week period.
  For evaluation of depressive symptoms was used the questionnaire PHQ-9 depression, which consists of nine items, including symptoms and attitudes whose intensity varies from zero to three, with 27 your score.
Sleep quality, evaluated by Pittsburgh Sleep Scale | At baseline and after a 15-week period.
  Sleep quality was assessed by Pittsburgh scale, consisting of 19 questions on the perception of oneself and five questions relating to the perception that the roommates of these individuals have about sleep the same. These questions are grouped into seven components, with score of zero to three.
Levels of sleep Obstructive Apnea, evaluated by Berlin Questionnaire (BQ) | At baseline and after a 15-week period.
  This questionnaire includes 10 items, organized in 3 categories related to snoring and apneas witnessed (5 items), daytime sleepiness (4 items) and high blood pressure (HTA) / obesity (1 item). Information on gender, age, height, weight, race neck circumference and is also requested. The determination of high or low risk to OSAS is based on responses in each category itens.
Physical activity levels, evaluated by International Physical Activity Questionnaire (IPAQ) - Short Form. | At baseline and after a 15-week period.
  The IPAQ short form asks about three specific types of activity undertaken in the three domains introduced above and sitting. The specific types of activity that are assessed are walking, moderate-intensity activities and vigorous intensity activities; frequency (measured in days per week) and duration (time per day) are collected separately for each specific type of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delevatti RS, Reichert T, Bracht CG, Lisboa SDC, Marson EC, Costa RR, Kanitz AC, Bones V, Stein R, Kruel LFM. Aquatic Aerobic and Combined Training in Management of Type 2 Diabetes: The Diabetes and Aquatic Training Study (DATS): A Randomized Clinical Trial. J Phys Act Health. 2022 Jul 28;19(8):578-587. doi: 10.1123/jpah.2022-0016. Print 2022 Aug 1. PMID 35902075
- [Derived] Delevatti RS, Kanitz AC, Bracht CG, Lisboa SDC, Marson EC, Reichert T, Bones V, Kruel LFM. Effects of 2 Models of Aquatic Exercise Training on Cardiorespiratory Responses of Patients With Type 2 Diabetes: The Diabetes and Aquatic Training Study-A Randomized Controlled Trial. J Phys Act Health. 2020 Sep 29;17(11):1091-1099. doi: 10.1123/jpah.2020-0236. PMID 32994381